CLINICAL TRIAL: NCT02424045
Title: A Phase II Trial of Bendamustine, Carboplatin and Dexamethasone (BCD) for Refractory or Relapsed Peripheral T-cell Lymphoma: BENCART Trial
Brief Title: Bendamustine, Carboplatin and Dexamethasone (BCD) for Refractory or Relapsed Peripheral T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Clinical Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-12-012
Record Dates: First submitted 2015-04-15; First posted 2015-04-22 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — Bendamustine Hydrochloride; Carboplatin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BCD chemotherapy (Other): All patients are scheduled to receive 2 cycles of three-weekly Bendamustine, carboplatin and dexamethasone combination chemotherapy(BCD Chemotherapy).
  D1,D2 Bendamustine 80mg/m2 IV over 30-60min D1 Carboplatin AUC 5.0 IV D1-4 Dexamethasone 40mg #2 PO or IV
  Interventions: Drug: BCD chemotherapy (Bendamustine, Carboplatin, Dexamethasone)

INTERVENTIONS:
Drug: BCD chemotherapy (Bendamustine, Carboplatin, Dexamethasone) — All patients are scheduled to receive 2 cycles of three-weekly BCD. After 2 cycles of BCD, if the patients with complete remission (CR) or partial remission (PR) would be eligible for autologous stem cell transplantation (ASCT), stem cell collection after 3rd cycle of BCD and high dose chemotherapy and ASCT will be conducted. While ineligible patients to ASCT with non-progressive disease after 2 cycles of BCD, will be given 4 additional courses of the BCD regimen.
  Other Names: BCD chemotherapy

SUMMARY:
BCD (Bendamustine, carboplatin and dexamethasone)chemotherapy regimen is proposed as the salvage treatment for relapsed or refractory PTCLs in this study protocol, which would be expected to show more promising clinical outcomes than that of bendamustine single therapy. Platinum combination with bendamustine is a theoretically ideal salvage regimen for the patients of PTCLs because these both agents are highly effective drugs in lymphoma treatment and have rare cross-resistance. Carboplatin was selected as a platinum agent for combination with bendamustine, which is a second generation platinum agent and has a less neurotoxicity than that of cisplatin, considering use for previously treated patients with vinc alkaloid agents.

In a prior phase I study of carboplatin in combination with bendamustine for previously untreated small cell lung cancer patients, the recommended dose for phase II studies was bendamustine 100 mg/m2 on day 1 and 2, carboplatin AUC 5 on day 1, respectively [16]. In consideration of previously treated subjects, however, the dose of bendamustine was decided on 80mg/m2 in this study protocol with concerning about the toxicities, especially to severe cytopenia.

Dexamethasone is one of the corticosteroids using a key drug for lymphoid malignancy and has a strong antiemetic effect. Therefore, dexamethasone could enhance the therapeutic efficacy and antiemetic effect, using with bendamustine and carboplatin.

DETAILED DESCRIPTION:
Peripheral T-cell lymphoma (PTCL) represents a heterogeneous group of nodal and extranodal mature T-cell lymphomas, which constitute about 5 - 10% of all non-Hodgkin lymphomas (NHLs) in Western countries compared to 20 - 30% of all lymphomas in the East Asia. The most common histologies include PTCL, not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), and anaplastic large cell lymphoma (ALCL) [3]. Most of these subtypes include a high percentage of patients with advanced disease stage, widespread dissemination and aggressive behavior. As a result, the prognosis of PTCL remains dismal, with the 5-year overall survival (OS) rate for many of these subtypes ranging between 25 and 45%, except for ALCL (ALK ), which demonstrates a better 5-year OS (70%) [4 - 6]. Thus, new therapeutic strategies are needed to improve the survival of patients with PTCL.

Current multiagent chemotherapeutic regimens for patients with PTCL are extrapolated mainly from therapeutic paradigms of B-cell lymphomas, with the cornerstone treatment being an anthracycline-containing regimen. Although some patients with PTCL can be cured with these approaches, relapsed and chemorefractory disease constitutes a significant clinical dilemma in the care of these patients [7]. At present, high dose chemotherapy with autologous stem cell support seems to offer potential curative treatment for those patients with relapsed PTCL who are responsive to salvage chemotherapy [8]. However, the majority of elderly patients with relapsed or refractory PTCL cannot benefit from high dose chemotherapy as a result of advanced age, significant comorbidities, poor functional status, toxicities from previous treatments and inherent chemoresistance [9]. Conventional salvage regimens have been mostly designed for younger or fitter populations, and can hardly be delivered to these elderly patients due to marked hematologic and non-hematologic toxicities, mainly involving renal and neurological functions [10]. Therefore, it is imperative that innovative salvage regimens based on drug combinations with increased efficacy and reduced toxicity be explored for the management of elderly patients with relapsed or refractory PTCLs.

BCD chemotherapy regimen is proposed as the salvage treatment for relapsed or refractory PTCLs in this study protocol, which would be expected to show more promising clinical outcomes than that of bendamustine single therapy. Platinum combination with bendamustine is a theoretically ideal salvage regimen for the patients of PTCLs because these both agents are highly effective drugs in lymphoma treatment and have rare cross-resistance. Carboplatin was selected as a platinum agent for combination with bendamustine, which is a second generation platinum agent and has a less neurotoxicity than that of cisplatin, considering use for previously treated patients with vinc alkaloid agents.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven aggressive T-cell Non-Hodgkin's lymphoma (NHL)
2. Age 18 -75 years
3. Ann Arbor stage II, III and IV (Appendix A)
4. Relapsed or refractory cases to previous treatments
5. Performance status (ECOG) ≤ 2 (Appendix B)
6. At least one or more bidimensionally measurable lesion(s)

   * ≥ 2 cm by conventional CT
   * ≥ 1 cm by spiral CT
   * skin lesion (photographs should be taken) ≥ 2 cm
   * measurable lesion by physical examination ≥ 2 cm
7. Cardiac ejection fraction ≥ 50 % as measured by MUGA or 2DECHO without clinically significant abnormalities
8. Adequate renal function: serum creatinine level < 2 mg/dL (177 μmol/L)
9. Adequate liver functions: Transaminase (AST/ALT) < 3 X upper normal value (or < 5 x ULN in the presence of DLBCL involvement of the liver), Bilirubin < 2 X upper normal value (or < 5 x ULN in the presence of PTCL involvement of the liver)
10. Adequate BM functions: hemoglobin ≥ 9 g/dL absolute neutrophil count (ANC) ≥ 1,500/μL and platelet count ≥ 75,000/μL, unless abnormalities are due to bone marrow involvement by lymphoma
11. A negative serum or urine pregnancy test prior to treatment must be available both for pre-menopausal women and for women who are < 1years after the onset of menopause.
12. Informed consent

Exclusion Criteria:

1. ALK-positive anaplastic large cell lymphoma and Sezary syndrome.
2. CNS or testis involvement.
3. Previously treated with the regimen containing bendamustine or platinum agents.
4. Any other malignancies within the past 5 years except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
5. Pregnant or lactating women, women of childbearing potential not employing adequate contraception
6. Other serious illness or medical conditions
7. Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry
8. History of significant neurologic or psychiatric disorders including dementia or seizures
9. Active uncontrolled infection (viral, bacterial or fungal infection)
10. Other serious medical illnesses
11. Known hypersensitivity to any of the study drugs or its ingredients
12. Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 3 years
  They should be classified as complete remission (CR), partial remission (PR), stable disease (SD), or progressive disease (PD) according to the Revised Response Criteria for Malignant Lymphoma

SECONDARY OUTCOMES:
Toxicity profiles (Adverse Events and Laboratory Results) | 3 years
  Toxicity profiles as measured by Adverse Events and Laboratory Results.The intensity of clinical adverse events will be graded according to the NCI CTCAE version 4.0.
Progression free survival | 3 years
  Time to disease progression is defined as the time from treatment start to the first recording of relapse or disease progression or death of any cause.
Overall survival | 3 years
  Duration of survival is defined as the time from treatment start to death of any cause or the date of last follow-up. Patients who are alive will be censored using the date at which they are last known to be alive.
Incidence of febrile neutropenia | 3 years

REFERENCES:
- [Derived] Park BB, Kim WS, Suh C, Hong JY, Yang DH, Lee WS, Do YR, Koh YI, Won JH, Kim MK, Jo JC, Hyun SY, Kim JA, Oh YH, Lee SS. A phase II trial of bendamustine, carboplatin, and dexamethasone for refractory or relapsed peripheral T-cell lymphoma (BENCART trial). Leuk Lymphoma. 2019 Dec;60(13):3251-3257. doi: 10.1080/10428194.2019.1622100. Epub 2019 Jun 6. PMID 31170847